CLINICAL TRIAL: NCT05519787
Title: A Retrospective, Observational, Monocenter, Study to Describe the Utilization and Overall Safety and Performance of POLYSITE®/SEESITE® Implantable Ports
Status: Completed | Type: Observational
Sponsor: Perouse Medical (Industry)
Collaborators: Eclevar Medtech (Industry)
Responsible Party: Sponsor
Other Study IDs: PSSS-2021-MONO
Record Dates: First submitted 2022-08-26; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Venous System; Venous Access; Chemotherapy; Antibiotics; Antiviral; Parenteral Nutrition; Transfusion Blood
MeSH Terms: conditions — Hyperphagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Central Veinous access devices' insertion — Medical doctor should complete a questionnaire with medical history or any important clinical data that could help for the selection of the location of the port and catheter placement. The insertion will be planned only by a surgeon, interventional radiologist, or anaesthesiologist in the surgery block.
  For the patient with a medical history of PICC line, PAC implantation, Central venous access device of any kind, or clinical risk of veinous compression (cervical or subclavian adenopathy, pelerine syndrome, mediastinal involvement…). An echo Doppler exam of the veinous cervical system is required before surgery. This exam should identify potential thrombosis that required a special treatment. It is important that the surgeon who will perform the device's insertion is aware of any history or risks of veinous thrombosis, stenosis, or phlebitis for the patient to avoid procedure's failure.

SUMMARY:
This study is a retrospective, observational, monocenter case series. The purpose of this study is to collect clinical data to describe the use of POLYSITE® and SEESITE® devices and verify overall safety and performance. This study is part of the Post-Market Clinical Follow-up (PMCF) activities of the PEROUSE MEDICAL manufacturer.

The primary data source for this study was patient's medical records from a French Hospital. The study population was defined as all patients who did receive POLYSITE® and SEESITE®. Data from a minimum of 50 patients were planned for the statistical review.

ELIGIBILITY:
Inclusion Criteria:

* Adult and pediatric population
* Patient who received the implantation of any POLYSITE® or SEESITE® implantable port referenced in the Annex 1 of the current protocol between 1st October 2016 and 31st December 2017

Exclusion Criteria:

* Patient who refused the data collection according to RGPD regulation applicable in France
* Patient who received the implantation of another device than those presented in Annex 1 of the current protocol.
* Patient who received the implantation of a POLYSITE® or SEESITE® implantable port after 31st December 2017

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population was defined in the protocol as all patients who did receive POLYSITE® or SEESITE® device between 1st October 2016 and 31 December 2017.
  Any patient who has disagreed with the collection of their personal data would be excluded from this study.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2022-05-19 (Actual); Study Completion 2022-05-19 (Actual)

PRIMARY OUTCOMES:
Identification of veins selected | 30 days
  insertion's location of the POLYSITE®/SEESITE® implantable port
rate of peri-operative complication | Peri-operative procedure
  number of complications between the implantation of the device and the first use (as example infections related to manipulation)

SECONDARY OUTCOMES:
type of treatments administered | 5 years
  chemotherapy, antibiotics, parenteral nutrition, other
Rate of procedural success | Peri-operative procedure
  correct placement and correct flow both confirmed by a radiological exam or an echography or an ECG.
short-term complication | 30 Days
  number of complications: infections, bleeding and hematoma, pneumothorax, hemothorax and pleural effusion, pain, and mechanical dysfunction (catheter fracture, occlusion, and port-pocket dehiscence, pinch-off, embolization, leak, port/catheter disconnection
rate of long-term complications | 5 years
  number of complications after 30 days of the implantation surgery up to the end of the follow-up: infections, inflammation, skin disorders, catheter-related venous thrombosis, mechanical dysfunction as occlusion/rupture/fracture/disconnection of the catheter, drug extravasation, mal-position, flip-over, migration, pinch-off.

CONTACTS AND LOCATIONS:
Locations (1):
- CHR d'Orléans, Orléans, France